CLINICAL TRIAL: NCT02832232
Title: Effectiveness of a Manual Specific Approach to the Suboccipital Area on Pain, Range of Motion, Disability and Clinical Significance of Changes on Patients With Chronic Mechanical Neck Pain and Rotation Deficit of the Upper Cervical Spine
Brief Title: Specific Manual Approach to the Suboccipital Area on Patients With Chronic Mechanical Neck Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P16/068
Record Dates: First submitted 2016-07-06; First posted 2016-07-14 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2016-05

CONDITIONS: Neck Pain
Keywords: Physiotherapy; Manual Therapy; Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mobilization Group (Experimental): translational dorsal glide mobilization technique grade III and Protocolized Physiotherapy
  Interventions: Other: translational dorsal glide mobilization technique grade III; Other: Control Group
- Maintained pressure Group (Experimental): pressure maintained suboccipital inhibition technique and Protocolized Physiotherapy
  Interventions: Other: pressure maintained suboccipital Inhibition technique; Other: Control Group
- Control Group (Other): Protocolized Physiotherapy
  Interventions: Other: Control Group

INTERVENTIONS:
Other: translational dorsal glide mobilization technique grade III — Translational dorsal glide mobilization technique grade III of the atlanto-occipital joint, it is a mobilization technique of Orthopedic Manual therapy according to Kaltenborn-Evjenth concept. The aim is to produce a dorsal glide of the occipital on the atlas, which will be held back by the therapist's hand, producing a stretch component of the suboccipital muscles.
  And Protocolized physiotherapeutic treatment: Three weeks of daily sessions (five a week) of stretching exercises, thermotherapy and postural education.
  Arms: Mobilization Group
Other: pressure maintained suboccipital Inhibition technique — Pressure maintained suboccipital Inhibition technique is aimed to inhibit the tone of the suboccipital muscles. Although some dorsal occipital glide is produced by the weight of the head itself, the main effect is on the muscles due to dorsally pressure is not added to the occipital.
  And Protocolized physiotherapeutic treatment: Three weeks of daily sessions (five a week) of stretching exercises, thermotherapy and postural education.
  Arms: Maintained pressure Group
Other: Control Group — Protocolized physiotherapeutic treatment: Three weeks of daily sessions (five a week) of stretching exercises, thermotherapy and postural education.

SUMMARY:
There are different inhibition suboccipital techniques, usually adjuvant of physiotherapy, for treatment of patients with chronic neck pain. In our clinical practice, a favorable effect is observed on patients with chronic neck pain, but there are no published studies evaluating the results of this techniques on pain, mobility and disability.

The objective of this trial is to evaluate if the suboccipital manual techniques, provides further improvement in pain intensity, neck disability, range of motion, on patients with chronic mechanical neck pain and rotation deficit of the upper cervical spine, being treated with physiotherapy. For this purpose, investigators conduct a double-blind (patient and evaluator) randomized controlled trial, in a Public Primary Care Center.

Seventy four subjects will be randomized (computer application) into three groups: Mobilization Group, Maintained pressure Group and Control Group. All the three groups receive the same protocolized physiotherapeutic treatment during three weeks and, additionally, the Mobilization Group receives six sessions (two sessions in a week during three weeks) of translational dorsal glide mobilization technique grade III of the atlanto-occipital joint and the Maintained pressure Group receives six sessions (two sessions in a week during three weeks) of pressure maintained suboccipital Inhibition technique. The Control Group receives the protocolized physiotherapeutic treatment only.

Pain intensity (VAS), Neck Disability Index (NDI), Range of motion (CROM), will be measured at baseline, after treatment period, and three months after discharge from treatment. After discharge for treatment the patient subjective opinion about their evolution will be collected through a Global Rating of Change (GROC) scale, and evaluation of headache disability (HIT-6).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic mechanical neck pain.
* Flexion-rotation test positive (less of 32 degrees or 10 degrees difference between the two sides)
* Sign the informed consent form.

Exclusion Criteria:

* Presenting one or more positive safety cervical test .
* Carriers of pacemaker or defibrillators.
* Previous history of severe trauma to the cervical region of the spine.
* Inflammatory arthritis.
* Inability to maintain supine position.
* Inability to tolerate flexion-rotation test
* Poor Language and communication skills making difficult to understand the informed consent.
* Pending litigation or legal claim.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain intensity | Baseline -3 weeks - 3 months
  Changes from Baseline in Pain intensity at 3 weeks and 3 months. Measure instrument: Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Changes in Neck disability | Baseline -3 weeks - 3 months
  Changes from Baseline in Neck disability at 3 weeks and 3 months. Measure instrument: Neck disability index questionnaire (NDI)
Changes in Range of motion | Baseline -3 weeks - 3 months
  Changes from Baseline in Range of Motion at 3 weeks and 3 months. Measure instrument: Cervical Range of Motion (CROM) device.
Patient perception of change at short term | 3 weeks after recruitment
  Measure instrument: Global Rating of Change scale (GROC-scale)
Patient perception of change at middle term | 3 weeks after discharge
  Measure instrument: Global Rating of Change scale (GROC-scale)
Headache disability at short term | 3 weeks after recruitment
  Measure instrument: Headache impact test (HIT-6)
Headache disability at middle term | 3 weeks after discharge
  Measure instrument: Headache impact test (HIT-6)

CONTACTS AND LOCATIONS:
Locations (1):
- Catalan Institut of Health - Sant Ildefons Rehabilitation Center, Cornellà de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Rueda V, Lopez-de-Celis C, Bueno-Gracia E, Rodriguez-Sanz J, Perez-Bellmunt A, Barra-Lopez ME, Hidalgo Garcia C. "Short- and mid-term effects of adding upper cervical manual therapy to a conventional physical therapy program in patients with chronic mechanical neck pain. Randomized controlled clinical trial.". Clin Rehabil. 2021 Mar;35(3):378-389. doi: 10.1177/0269215520965054. Epub 2020 Oct 19. PMID 33076707
- [Derived] Gonzalez Rueda V, Lopez de Celis C, Barra Lopez ME, Carrasco Uribarren A, Castillo Tomas S, Hidalgo Garcia C. Effectiveness of a specific manual approach to the suboccipital region in patients with chronic mechanical neck pain and rotation deficit in the upper cervical spine: study protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2017 Sep 5;18(1):384. doi: 10.1186/s12891-017-1744-5. PMID 28870191